CLINICAL TRIAL: NCT02997592
Title: Evaluation of the SpinCare™ System in the Treatment of Partial Thickness Burns - A Prospective Single Arm, Safety and Efficacy, Open Labeled Multi-center Study
Brief Title: Evaluation of the SpinCare™ System in the Treatment of Partial Thickness Burns
Acronym: SPINCARE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanomedic Technologies Ltd. (Industry)
Responsible Party: Sponsor
Organization: Nicast Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP0009
Record Dates: First submitted 2016-11-22; First posted 2016-12-20 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Partial Thickness Burn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SpinCare (Experimental): Patients with partial thickness burns treated with the SpinCare System
  Interventions: Device: SpinCare

INTERVENTIONS:
Device: SpinCare — The burn wound is treated using the SpinCare Systen

SUMMARY:
Evaluation of the SpinCare™ System in the Treatment of Partial Thickness Burns. A prospective, single arm, safety and efficacy, open labeled multi-center study

DETAILED DESCRIPTION:
The SpinCare is an electrospinning portable device intended for the external treatment of burns and wounds. The SpinCare is the first made on the spot, bed side, and completely personalized dressing system; with excellent coverage of all size, shapes and difficult contours. The nano-fibrous dressing mimics the structure of natural body tissue and creates excellent medium for tissue repair and healing.

The objective of this study is to evaluate the performance, safety and efficacy of the SpinCare System in the treatment of superficial to intermediate partial thickness burns.

The study included 3 sites. Adult patients with superficial to intermediate partial thickness burns (second degree superficial to intermediate) of up to 10% TBSA (Total Body Surface Area); with an independent burn of up to 5% TBSA.

A prospective single arm, safety and efficacy, open labeled, multi-center study for the treatment of partial thickness burn wounds not considered for surgery using the SpinCare System.

44 patients enrolled in the study.

Endpoints:

* Wound healing and re-epithelialization on day 21.
* The burn will be considered healed when at least 95% of the total area is re-epithelialized and no scabs exist.

  * Ease of use
  * At postoperative days 7, 14, 21
* Dermal safety assessed by Draize Score
* Visual estimate of wound healing and re-epithelialization
* Pain
* Infection
* Itching

  * Itching and scar quality at 3 and 6 months
  * Itching and scar quality at 12 months (optional)
  * Device related adverse events

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old at enrolment. Both genders.
* The patient has partial thickness burn wounds (second degree superficial to intermediate) of up to 10% TBSA; of which the target wound for treatment is of up to 5% TBSA or up to 300cm2.
* Presenting at the emergency room within the first 24-48 hours post-injury.
* Patient's wound is defined as a partial thickness burn for conservative treatment (superficial to intermediate second degree).
* Patient underwent cleansing/debridement of initial burn before applying the dressing
* The patient is able and willing to comply with study procedures and give written informed consent prior to enrollment in the study

Exclusion Criteria:

* Any known or suspected systemic infection
* Any known sensitivity to components/products used in this study
* Any active, uncontrolled, progressive or untreated malignancy
* Use of penicillamine, corticosteroid or immunosuppressive medication within two months prior to enrollment or who is likely to be prescribed these medications or any other medications known to adversely affect wound healing during study participation
* Major uncontrolled systemic disorders such as hepatic, renal, neurologic, or endocrinologic disorders
* Major dermatological disorders such as: psoriasis, pemphigus, Steven Johnson, etc.
* Patients with burns larger than 10% TBSA
* Patients with burns up to 10% TBSA but no target wound of up to 5% TBSA or up to 300cm2
* Patients suffering from electrical or chemical burns.
* Patients suffering from frostbites.
* Patients suffering from burn wounds that are third degree or full thickness.
* Patients suffering from burn wounds in the head, neck or genital areas
* Female patients who are pregnant or nursing
* Psychiatric patient.
* Soldiers
* Participation in another clinical trial within 30 days prior to the Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Burn wound healing | 21 days
  Wound healing and re-epithelialization on day 21. The burn will be considered healed when at least 95% of the total area is re-epithelialized and no scabs exist.

SECONDARY OUTCOMES:
Dermal safety test (erythema and edema) | Every time the SpinCare dressing is delivered up to 21 days after initial dressing
  Dermal safety will be assessed by Draize score including signs of erythema and edema.
Pain as assessed by VAS | 21 days
  Pain will be assessed at rest, during dressing application (when applicable) and during dressing removal (when applicable) using VAS (Visual Analog Scale) scale.
Number of participants having an infection at the burn wound. | Up to 21 days after initial application of the dressing
  If infection is suspected clinically, a swab will be taken for microbiological examination and the patient will be treated according to the medical center's standard practice.
Ease of use | Every time the SpinCare is used up to 21 days after initial application of the dressing
  ease of applying and removing the dressing will be evaluated using 0-5 numerical rating scale (NRS).

CONTACTS AND LOCATIONS:
Overall Officials: Moti Harats, Dr, Principal Investigator — Sheba Medical Center
Locations (3):
- Israel (3):
  - Rambam Medical Center, Haifa
  - Burn Unit, Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No